CLINICAL TRIAL: NCT01788111
Title: Occurrence, Diagnosis and Treatment of Neck and Back Pain in Helicopter Pilots.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUS-ID 294; 2010/2254/REK vest (Other: REK / Norway)
Record Dates: First submitted 2013-02-05; First posted 2013-02-11 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2019-12

CONDITIONS: Low Back Pain; Neck Pain; Muscular Atrophy
MeSH Terms: conditions — Low Back Pain; Neck Pain; Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low back exercises 1 (Experimental): Specific low back extensor exercises in special training bench
  Interventions: Other: Low back exercises 1
- Low back exercise 2 (Active Comparator): Traditional low back exercises.
  Interventions: Other: Low back exercise 2

INTERVENTIONS:
Other: Low back exercises 1 — Excentric / concentric extension type exercises
  Arms: Low back exercises 1
Other: Low back exercise 2 — Traditional low back training
  Arms: Low back exercise 2

SUMMARY:
The purpose of this project is to investigate the occurrence of neck and back pain in a population of commercial helicopter pilots, and investigate factors related to the profession that can cause these problems. The project has a biological approach assessing the supporting and stabilizing muscles (multifidus) in pilots with chronic back and neck ailments. Pilots with low back problems are invited to a controlled intervention trial to investigate whether one can achieve improved spinal health with a rigid training régime. Primary trial outcome is improved neck and back multifidus muscles pathology and function as assessed by the extent of fat infiltration -as visualized on MRI - and the volume and ability of the lumbar multifidus muscles to contract as shown with ultrasound. The perceived effect on spinal health with sick leave frequency is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Pilots must experience low back pain in at least 1 of 3 flights or
* Pilots must have at least 2 episodes of low back pain of at least 24 hours duration over the last 12 months. Each episode is separated with at least one painfree month before and after each episode, or
* Pilots may have had more than 3 sick leaves due to low back pain over the last 5 years

Exclusion Criteria:

* contraindications for physical training/activity

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 325 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Multifidus muscle fat infiltration (% of muscle volume). | one year
  Primary trial outcome is improved neck and back multifidus muscles pathology and function as assessed by the extent of fat infiltration as visualized on MRI (% of muscle volume).Change from baseline at 12 months.

SECONDARY OUTCOMES:
Lumbar multifidus muscles contractability. | Two years
  Volume and ability of the lumbar multifidus muscles to contract as shown with ultrasound (% of expansion during reflex activation)Change from baseline at 3,6,9,12 and 24 months.

OTHER OUTCOMES:
Number and duration of sick leaves amongst helicopter pilots | Two years
  Effect on spinal health with sick leave frequency in helicopter pilots. Change from baseline in numbers and duration compared to previous years statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Jan P Larsen, Prof.Dr.Med, Study Chair — Research Dep. Stavanger University Hospital
Locations (1):
- Research Dep. Stavanger University Hospital Armauer Hansens vei 20 PB 8100 4068 Stavanger, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen K, Baardsen R, Dalen I, Larsen JP. Recurrent and Transient Spinal Pain Among Commercial Helicopter Pilots. Aerosp Med Hum Perform. 2015 Nov;86(11):962-9. doi: 10.3357/AMHP.4237.2015. PMID 26564761
- [Background] Andersen K, Baardsen R, Haga H, Due G, Dalen I, et al. (2017) Transient Low Back Pain among Helicopter Pilots; Imaging and Lumbar Trunk Muscular Endurance. J Phys Med Rehabil Disabil 3: 021
- [Background] Andersen K, Baardsen R, Dalen I, Larsen JP. Impact of exercise programs among helicopter pilots with transient LBP. BMC Musculoskelet Disord. 2017 Jun 20;18(1):269. doi: 10.1186/s12891-017-1631-0. PMID 28633669
- [Background] Andersen K, Baardsen R, Dalen I, Larsen JP. Long-term effects of exercise programs among helicopter pilots with flying related LBP. J Back Musculoskelet Rehabil. 2018 Feb 6;31(1):1-13. doi: 10.3233/BMR-170897. PMID 29278872